CLINICAL TRIAL: NCT01172210
Title: Examining Common Substrates of Eating and Alcohol Use Disorders
Status: Completed | Type: Observational
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Sponsor
Other Study IDs: #5973/6951R
Record Dates: First submitted 2010-07-28; First posted 2010-07-29 (Estimated); Last update posted 2014-08-21 (Estimated); Status verified 2013-04

CONDITIONS: Bulimia Nervosa; Alcohol Use Disorders
MeSH Terms: conditions — Bulimia Nervosa; Alcoholism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Bulimia Nervosa
- Bulimia Nervosa w/ Alcohol Use Disorder
- Healthy Controls

SUMMARY:
A substantial percentage of individuals with bulimia nervosa (BN) also meet criteria for a co-occurring substance use disorder, such as alcohol abuse or dependence; however, research examining this sub-group of patients with BN is limited. Understanding characteristics common to both eating and alcohol use disorders may enhance understanding of the mechanisms that could contribute to the co-occurrence and perpetuation of these disorders. Individuals with BN and alcohol use disorders appear to share some behavioral traits, and therefore, the primary aim of the current study is to compare patients with BN with and without an alcohol use disorder and normal controls on measures assessing an individual's mood and ability to perform certain tasks. Participants will be asked to complete computer-administered and paper-and-pencil assessments and two laboratory test meals on separate days. By probing the underpinnings of BN and alcohol use disorders, the investigators can determine whether these disorders have a shared diathesis, which will lay an essential foundation for future research to examine biological and genetic correlates of these disorders. Finally, as little is known about the treatment of patients with BN and a co-occurring alcohol use disorder, an exploratory aim of the current study is evaluate the suitability and efficacy of a 20-session cognitive-behavioral treatment (CBT) addressing both bulimic symptoms and alcohol use.

DETAILED DESCRIPTION:
A substantial percentage of individuals with bulimia nervosa (BN) also meet criteria for a co-occurring substance use disorder, such as alcohol abuse or dependence; however, research examining this sub-group of patients with BN is limited. Understanding characteristics common to both eating and alcohol use disorders may enhance our understanding of the mechanisms that could contribute to the co-occurrence and perpetuation of these disorders. The primary aim of the current study is to compare patients with BN with and without an alcohol use disorder and normal controls on computer-administered and paper-and-pencil assessments and in two laboratory test meals (a binge meal and a normal meal) on separate days. Participants will also complete self-report and interview measures of eating disorder symptoms and alcohol consumption. By probing the underpinnings of BN and alcohol use disorders, we can determine whether these disorders have a shared diathesis, which will lay an essential foundation for future research to examine biological and genetic correlates of these disorders. Finally, as little is known about the treatment of patients with BN and a co occurring alcohol use disorder, an exploratory aim of the current study is to evaluate the suitability and efficacy of a 20-session cognitive-behavioral treatment (CBT) addressing both bulimic symptoms and alcohol use.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-45
* Diagnosis of bulimia nervosa with or without a co-occurring alcohol use disorder
* English speaking
* Weight above 80% of ideal

Exclusion Criteria:

* Other significant psychiatric conditions requiring treatment or a significant medical condition
* Pregnancy
* Current use of psychotropic medication
* History of neurological disorder (e.g., dementia, stroke seizure)
* Food allergy to items in the lunch buffet
* Positive urine drug screen
* Current or post eating disorder diagnosis or history of binge eating or vomiting
* Current or past alcohol or substance abuse or dependence

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participants who call the main clinic line at the Eating Disorders Research Unit at NYSPI/CUMC.
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2009-07; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Eating Behavior | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Robyn Sysko, Ph.D., Principal Investigator — New York State Psychiatric Institute
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

REFERENCES:
- See also: Related Info — http://columbiaeatingdisorders.org/